CLINICAL TRIAL: NCT06723418
Title: Development and Validation of a New Paediatric Inflammatory Bowel Disease NUTrition Risk Score (PIBD-NUTS)
Acronym: PIBD-NUTS
Status: Recruiting | Type: Observational
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Konstantinos Gerasimidis, Professor of Clinical Nutrition, University of Glasgow
Other Study IDs: PIBD-NUTS
Record Dates: First submitted 2024-12-02; First posted 2024-12-09 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Inflammatory Bowel Diseases (IBD); Crohns Disease; Ulcerative Colitis (UC)
Keywords: Ulcerative colitis; Crohns disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric patients with Inflammatory Bowel Disease (Crohns disease & ulcerative colitis)
  Interventions: Other: Malnutriton Screening Tool (PYMS)

INTERVENTIONS:
Other: Malnutriton Screening Tool (PYMS) — In a pilot implementation study, PYMS will be used on children with IBD attending the outpatient and inpatient hospital clinics

SUMMARY:
Children with inflammatory bowel disease (IBD) including both Crohn's disease (CD) and ulcerative colitis (UC) can be at high risk of developing malnutrition due to the nature of their condition. It is also believed that some children with IBD, in need of nutritional care, are not identified quickly by their healthcare professionals. This may negatively affect their nutrition, disease progression and general well-being. Hence, it has been proposed that nutritional screening tools or scores (NSTs) should be used to promptly identify children needing further dietetic review and input. Although there are a few NSTs for generic use in sick children at hospital admission, NSTs or scores to use for children with IBD are currently missing. In this study, we would like to test the performance of an existing tool that is routinely used for all sick children at hospital admission (The Paediatric Yorkhill Malnutrition Score or PYMS)(5) and test whether PYMS can detect children with IBD who are at risk of malnutrition. If PYMS doesn't work well, we will develop a specific tool for children with IBD (The Paediatric IBD Nutrition Score or PIBD-NUTS).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with either Crohn's disease or ulcerative colitis between the ages of (4-18 years)

Exclusion Criteria:

* Pediatric patients with IBDU

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All IBD (Crohns disease & ulcerative colitis) patients (4-18 years) either admitted to hospital, or visiting their gastroenterologist's outpatient clinic for routine visits are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
the performance of an existing nutritional screening tool (PYMS) in paediatric IBD patients at different international settings. | 1 year
  The primary outcome measure for our study is to evaluate the performance of an existing nutritional screening tool, the Paediatric Yorkhill Malnutrition Score (PYMS), specifically in pediatric IBD patients across various international settings. We aim to assess its diagnostic accuracy by examining sensitivity and specificity.

CONTACTS AND LOCATIONS:
Locations (8):
- Salzburg University Hospital, Salzburg, Austria
- Children's Hospital Zagreb, Zagreb, Croatia
- University of Giessen, Giessen, Germany
- Erasmus MC university medical centre, Rotterdam, Netherlands
- The Children's Memorial Health Institute, Warsaw, Poland
- United Kingdom (3):
  - University Hospital Bristol and Weston, Bristol
  - Royal Hospital for Children and Young People, Edinburgh
  - Great Ormond Street Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerasimidis K, Keane O, Macleod I, Flynn DM, Wright CM. A four-stage evaluation of the Paediatric Yorkhill Malnutrition Score in a tertiary paediatric hospital and a district general hospital. Br J Nutr. 2010 Sep;104(5):751-6. doi: 10.1017/S0007114510001121. Epub 2010 Apr 19. PMID 20398432
- [Background] Gerasimidis K, Macleod I, Maclean A, Buchanan E, McGrogan P, Swinbank I, McAuley M, Wright CM, Flynn DM. Performance of the novel Paediatric Yorkhill Malnutrition Score (PYMS) in hospital practice. Clin Nutr. 2011 Aug;30(4):430-5. doi: 10.1016/j.clnu.2011.01.015. Epub 2011 Mar 9. PMID 21388725
- [Background] Ng SC, Shi HY, Hamidi N, Underwood FE, Tang W, Benchimol EI, Panaccione R, Ghosh S, Wu JCY, Chan FKL, Sung JJY, Kaplan GG. Worldwide incidence and prevalence of inflammatory bowel disease in the 21st century: a systematic review of population-based studies. Lancet. 2017 Dec 23;390(10114):2769-2778. doi: 10.1016/S0140-6736(17)32448-0. Epub 2017 Oct 16. PMID 29050646
- [Background] Hulst JM, Huysentruyt K, Gerasimidis K, Shamir R, Koletzko B, Chourdakis M, Fewtrell M, Joosten KF; Special Interest Group Clinical Malnutrition of ESPGHAN. A Practical Approach to Identifying Pediatric Disease-Associated Undernutrition: A Position Statement from the ESPGHAN Special Interest Group on Clinical Malnutrition. J Pediatr Gastroenterol Nutr. 2022 May 1;74(5):693-705. doi: 10.1097/MPG.0000000000003437. Epub 2022 Mar 3. PMID 35258497
- [Background] Gerasimidis K, McGrogan P, Edwards CA. The aetiology and impact of malnutrition in paediatric inflammatory bowel disease. J Hum Nutr Diet. 2011 Aug;24(4):313-26. doi: 10.1111/j.1365-277X.2011.01171.x. Epub 2011 May 13. PMID 21564345